CLINICAL TRIAL: NCT06872684
Title: Safety and Efficacy of Endovascular Treatment of Intracranial Aneurysms With Surpass Elite With GUARDian Flow Diverter
Brief Title: Safety and Efficacy of Endovascular Treatment of Intracranial Aneurysms With Surpass Elite With GUARDian Flow Diverter (GUARD)
Acronym: GUARD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDM10001836
Record Dates: First submitted 2025-02-27; First posted 2025-03-12 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Aneurysm; Aneurysm, Intracranial
Keywords: Saccular Aneurysm; Fusiform Aneurysm; Unruptured Aneurysm; Flow Diverter
MeSH Terms: conditions — Aneurysm; Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Surpass Elite with Guardian Flow Diverter (Experimental): This is a prospective single arm study in which all subjects who present for Surpass Elite with Guardian flow diverter implantation, provide informed consent, and meet inclusion/exclusion criteria may receive treatment.
  Interventions: Device: Surpass Elite with Guardian Flow Diverter System

INTERVENTIONS:
Device: Surpass Elite with Guardian Flow Diverter System — The Surpass Elite with Guardian Flow Diverter System is indicated for use in the endovascular treatment of adults (age 18 or above) with unruptured wide-neck saccular or fusiform intracranial aneurysms arising from a parent vessel with a diameter ≥ 3.0 millimeter (mm) and ≤ 6.0 mm and located on the Internal Carotid Artery (ICA) or its branches.

SUMMARY:
The objective of the Safety and Efficacy of Endovascular Treatment of Intracranial Aneurysms with Surpass Elite with GUARDian Flow Diverter (GUARD) trial is to evaluate the safety and efficacy of the Surpass Elite with Guardian Flow Diverter System (FDS) in the treatment of unruptured, wide-neck saccular or fusiform, intracranial aneurysms (IAs) located on the internal carotid artery (ICA) or its branches.

DETAILED DESCRIPTION:
The Surpass Elite with Guardian Flow Diverter System is indicated for use in the endovascular treatment of adults (age 18 or above) with unruptured wide-neck saccular or fusiform intracranial aneurysms arising from a parent vessel with a diameter ≥ 3.0 millimeters (mm) and ≤ 6.0 mm and located on the ICA or its branches.

ELIGIBILITY:
Inclusion Criteria:

1. Age is ≥18 and ≤80 years at the time of consent
2. Has a single unruptured target intracranial aneurysm (IA) of any size with the following characteristics:

   1. Is located on the internal carotid artery or its branches
   2. Has a wide neck (wide neck typically defined as neck width ≥ 4 millimeter (mm), or dome to neck ratio ≤ 2.0) or no discernible neck
   3. Aneurysm is either saccular or fusiform in nature
3. Has a parent vessel diameter ≥ 3.0 mm to ≤ 6.0 mm at the largest diameter
4. There is documented risk-benefit of endovascular treatment that outweighs the risks of intracranial aneurysm rupture during the subject's expected lifetime if left untreated.

Exclusion Criteria:

1. Has an extradural target aneurysm
2. Has a target aneurysm in the posterior circulation
3. Perforator or branch vessel, inclusive of the posterior communicating artery, arises from the target aneurysm body or neck (branches or arteries must arise or connect from the parent vessel separate from the aneurysm or neck to not be excluded from trial)
4. Has a true bifurcation aneurysm, defined as an aneurysm (saccular or non-saccular) located at a point of vessel bifurcation
5. Has vessel characteristics, such as severe tortuosity (cavernous Internal Carotid Artery (cICA) Type IV1), stenosis (>70%), or morphology that would preclude safe endovascular access or proper deployment of the trial device to the target aneurysm
6. Received previous treatment for the target aneurysm or parent artery where it would interfere with the placement or proper apposition of the device
7. Has a medical contraindication to trial or procedure related antiplatelet medications (aspirin, clopidogrel/Plavix, ticagrelor, and heparin), local or general anesthesia, or life-threatening allergy to contrast dye
8. Has a known severe allergy to nickel, chromium cobalt, tungsten, or platinum
9. Patients with heparin hypersensitivity, including patients with a previous incident of Heparin-Induced Thrombocytopenia (HIT).
10. Modified Rankin Score (mRS) assessment is ≥ 3 at pre-procedure exam
11. Presence of unstable neurological deficit (i.e., worsening of clinical condition in the last 30 days prior to the index procedure)
12. Subarachnoid hemorrhage occurred within 30 days prior to the index procedure
13. Major surgery (including previous intracranial implant) either occurred within 30 days prior to the index procedure date or is planned to occur within 120 days following the index procedure date
14. Has more than one intracranial aneurysm (IA) that requires treatment within 12 months after the index procedure
15. Received previous intracranial implant associated with the symptomatic or vascular distribution within the past 84 days prior to treatment date
16. Chronic anticoagulation therapy is ongoing or known coagulopathy exists
17. Has atrial fibrillation with or without pacemaker.
18. Has other known serious concurrent medical conditions such as cardiovascular disease (including recent myocardial infarction [<12 weeks], symptomatic congestive heart failure, or carotid stenosis), kidney failure (>2.0 mg/dl serum creatinine), pulmonary disease, uncontrolled diabetes, progressive neurologic disorders, terminal cancer, vasculitis, high risk of ischemic stroke or recent stroke
19. Has acute life-threatening illness (e.g., acute kidney or heart failure) other than the neurological disease to be treated in this trial
20. Evidence of active infection at the time of treatment
21. Life expectancy is less than 5 years due to other illness or condition (in addition to an intracranial aneurysm)
22. Unable to comply with the trial follow up requirements due to conditions such as dementia or psychiatric problems, active substance abuse, or history of non-compliance with medical advice, as determined by the investigator
23. Pregnant or breast- feeding women or women who wish to become pregnant during the length of trial participation
24. Presence of intracranial mass (tumor, except meningioma, abscess, or other infection), non-treated arteriovenous malformation (AVM) in the territory of the target aneurysm
25. Enrollment in another study involving an investigational product that could confound the outcomes of this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
The primary safety endpoint: Number of subjects with neurologic death or major ipsilateral stroke through 12 months as adjudicated by an independent Clinical Events Committee (CEC). | 12 month ± 3 months
  Neurological death defined as stroke-related death and related to the vascular territory associated with target aneurysm treatment. Major ipsilateral stroke defined as a stroke with an increase in National Institutes of Health Stroke Scale (NIHSS) score ≥ 4 points persisting ≥ 24 hours and related to the vascular territory associated with target aneurysm treatment.
The primary efficacy endpoint: Number of subjects with 100% occlusion of the target aneurysm without significant parent artery stenosis, and with no target aneurysm retreatment through the 12-month follow-up visit timepoint. | 12 month ± 3 months
  The primary efficacy endpoint is a composite of 100% occlusion (Raymond-Roy Class 1, complete occlusion) of the target aneurysm without significant parent artery stenosis (significant parent artery stenosis is defined as > 50% stenosis, per independent core lab assessment of digital subtraction angiography [DSA] images acquired at 12 months [± 90 days] post-procedure), and with no target aneurysm retreatment through the 12-month follow-up visit timepoint.

SECONDARY OUTCOMES:
Secondary Safety Endpoint #1: Number of subjects with neurological death or disabling stroke as adjudicated by an independent Clinical Events Committee (CEC). | 12 month ± 3 months, 36 month ± 3 months, and 60 month ± 3 months if FDA grants Premarket approval (PMA) of the Surpass Elite with Guardian Flow Diverter System
  Neurological death defined as stroke-related death and related to the vascular territory associated with target aneurysm treatment. Disabling stroke defined as stroke related to the vascular territory associated with target aneurysm treatment that results in a modified Rankin Score (mRS) score ≥ 3, as assessed by an independent qualified (certified or with documented qualification per institution standard of care) assessor at a minimum of 90 days post stroke event.
  The number of subjects with neurological deaths or disabling strokes as adjudicated by an independent Clinical Events Committee (CEC) will be analyzed.
Secondary Safety Endpoint #2: Number of subjects with stroke related to the vascular territory associated with target aneurysm treatment as adjudicated by an independent Clinical Events Committee (CEC). | 12 month ± 3 months, 36 month ± 3 months, and 60 month ± 3 months if FDA grants Premarket approval (PMA) of the Surpass Elite with Guardian Flow Diverter System
  The number of subjects with strokes related to the vascular territory associated with target aneurysm treatment as adjudicated by an independent Clinical Events Committee (CEC) will be analyzed.
Secondary Safety Endpoint #3: Number of subjects with combined stroke and transient ischemic attack (TIA) events as adjudicated by a CEC | 12 month ± 3 months, 36 month ± 3 months, and 60 month ± 3 months if FDA grants Premarket approval (PMA) of the Surpass Elite with Guardian Flow Diverter System
  The number of subjects with combined stroke and transient ischemic attack (TIA) events as adjudicated by an independent Clinical Events Committee (CEC) will be analyzed
Secondary Efficacy Endpoint #1: Number of subjects with 100% occlusion (Raymond-Roy Class 1, complete occlusion) of the target aneurysm at follow-up visits | 12 month ± 3 months, 36 month ± 3 months, and 60 month ± 3 months if FDA grants Premarket approval (PMA) of the Surpass Elite with Guardian Flow Diverter System
  The number of subjects with 100% occlusion (Raymond-Roy Class 1, complete occlusion) of the target aneurysm at follow-up visits, per independent core lab assessment of DSA images will be analyzed
Secondary Efficacy Endpoint #2: Number of subjects with 100% occlusion of the target aneurysm at follow-up visits, per independent core lab assessment of any images (including but not limited to MRA and CTA) | 12 month ± 3 months, 36 month ± 3 months, and 60 month ± 3 months if FDA grants Premarket approval (PMA) of the Surpass Elite with Guardian Flow Diverter System
  100% occlusion (Raymond-Roy Class 1, complete occlusion) of the target aneurysm at follow-up visits, per independent core lab assessment of any images (including but not limited to MRA and CTA)
Secondary Efficacy Endpoint #3: Number of subjects with significant (> 50% stenosis) parent artery stenosis as determined by independent core lab post-procedure | 12 month ± 3 months, 36 month ± 3 months, and 60 month ± 3 months if FDA grants Premarket approval (PMA) of the Surpass Elite with Guardian Flow Diverter System
  The number of subjects with significant (> 50% stenosis) parent artery stenosis as determined by independent core lab post-procedure will be analyzed
Secondary Efficacy Endpoint #4: Number of subjects with target aneurysm retreatment. | 12 month ± 3 months, 36 month ± 3 months, and 60 month ± 3 months if FDA grants Premarket approval (PMA) of the Surpass Elite with Guardian Flow Diverter System
  The number of subjects with target aneurysm retreatment will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Coon, MD, Principal Investigator — Carondelet at St. Joesphs; David Fiorella, MD, Principal Investigator — Stony Brook University
Locations (3):
- United States (3):
  - Carondelet St. Joseph's Hospital, Tucson, Arizona
  - University of California Davis Health, Davis, California
  - Lahey Hospital and Medical Center, Burlington, Massachusetts